CLINICAL TRIAL: NCT01031030
Title: Adjuvant Treatment of Biologically Aggressive Breast Cancer (N-,N+1,3): Controlled Clinical Study
Brief Title: Cyclophosphamide, Methotrexate, and Fluorouracil, With or Without Epirubicin Hydrochloride, in Treating Women Who Have Undergone Surgery for Breast Cancer (Group III Closed to New Patients as of 12/7/2009)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: IRST-IBIS-03; CDR0000661068 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Epirubicin; Fluorouracil; Methotrexate; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: methotrexate
Other: laboratory biomarker analysis
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, methotrexate, fluorouracil, and epirubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving cyclophosphamide together with methotrexate and fluorouracil before, after, or without epirubicin hydrochloride is more effective in treating patients with breast cancer that can be removed by surgery.

PURPOSE: This randomized phase III trial is comparing three regimens of cyclophosphamide given together with methotrexate and fluorouracil, with or without epirubicin hydrochloride, to see how well it works in treating women who have undergone surgery for breast cancer. (Group III was closed to new patients as of 12/7/2009.)

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the impact of adjuvant chemotherapy comprising epirubicin hydrochloride followed by cyclophosphamide, methotrexate, and fluorouracil versus cyclophosphamide, methotrexate, and fluorouracil followed by epirubicin hydrochloride versus cyclophosphamide, methotrexate, and fluorouracil on overall survival of patients with biologically aggressive, resectable, node-negative or node-positive breast cancer.

Secondary

* To assess the disease-free survival and patterns of relapse in these patients.
* To assess the tolerance to and toxicity of treatment in these patients.
* To determine the quality of life of these patients.
* To verify the effectiveness of these treatments in different subgroups of patients.
* To collect, retrospectively, information on the expression of tumor suppressor gene p53, oncogene c-erbB-2, and bcl-2 protein involved in apoptosis. (exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to center, lymph node status (N0 vs N1-3), and estrogen receptor status (negative vs positive). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Beginning 4-6 weeks following surgery, patients receive epirubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive cyclophosphamide IV, methotrexate IV, and fluorouracil IV on days 1-8. Treatment repeats every 4 weeks for 4 courses.
* Arm II: Beginning 4-6 weeks following surgery, patients receive cyclophosphamide IV, methotrexate IV, and fluorouracil IV on days 1-8. Treatment repeats every 4 weeks for 4 courses. Patients then receive epirubicin hydrochloride IV on day 1. Treatment repeats every 3 weeks for 4 courses.
* Arm III (closed to accrual as of 12/7/2009): Beginning 4-6 weeks following surgery, patients receive cyclophosphamide IV, methotrexate IV, and fluorouracil IV on days 1-8. Treatment repeats every 4 weeks for 6 courses.

Patients with estrogen receptor-positive disease receive tamoxifen daily for 5 years after completing chemotherapy.

After completion of study therapy, patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Underwent radical mastectomy, guadrantectomy, or tumorectomy with axillary node dissection within the past 4-6 weeks
  * Biologically aggressive disease
  * At least 10 lymph nodes removed

    * Node-negative (> 1 cm, or > 2 cm if histology is favorable, esp. tubular carcinoma and/or prevalent intraductal component > 50%) tumors OR node-positive (1-3) tumors, meeting the following criteria:

      * High thymidine-labeling index (> 3%)
      * Poorly differentiated tumor (grade III)
      * High S-phase fraction (> 10% by flow cytometry)
      * High Ki67/MIB1 expression (< 20%)
* No bilateral breast cancer
* No T4a, inoperable T4b, T4c, or T4d disease
* Any estrogen receptor status (positive, negative, unknown)
* No distant metastases

PATIENT CHARACTERISTICS:

* Any menopause status
* WBC ≥ 3,500/mL
* ANC ≥ 1,500/mL
* Platelet count ≥ 120,000/mL
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 mg/mL
* Bilirubin ≤ 1.5 times ULN
* Not pregnant
* Geographically accessible for follow-up
* No prior breast cancer and/or other cancer except for carcinoma in situ of the cervix or basal cell skin cancer treated with radical intent
* No significant alterations in cardiovascular function
* No serious psychiatric disorders
* No impaired renal or liver function

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1997-11; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Disease-free survival
Toxicity
Quality of life
Efficacy in subgroups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Dino Amadori, MD, Principal Investigator — Morgagni-Pierantoni Ospedale

REFERENCES:
- [Derived] Farolfi A, Scarpi E, Rocca A, Mangia A, Biglia N, Gianni L, Tienghi A, Valerio MR, Gasparini G, Amaducci L, Faedi M, Baldini E, Rubagotti A, Maltoni R, Paradiso A, Amadori D. Time to initiation of adjuvant chemotherapy in patients with rapidly proliferating early breast cancer. Eur J Cancer. 2015 Sep;51(14):1874-81. doi: 10.1016/j.ejca.2015.07.003. Epub 2015 Jul 20. PMID 26206258